CLINICAL TRIAL: NCT02401269
Title: Cardiovascular Risk in HIV Patients on Antiretroviral Therapy Therapy: The MHEART Study
Acronym: MHEART
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); University of North Carolina (Other)
Responsible Party: Principal Investigator, Anil Purohit, MD, Cardiology Fellow, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO14040373
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Cardiovascular Disease Risk in HIV Patients; Endothelial Function
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspirin (Experimental): Aspirin 325mg daily
  Interventions: Drug: Aspirin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin
  Arms: Aspirin
Drug: Placebo
  Arms: Placebo

SUMMARY:
CVD accounts for 15% of all deaths in Malawi. Both HIV and ART are risk factors for CVD through direct toxic and inflammatory cardiovascular effects. (44,45). At the moment, one out of every 10 Malawian is HIV positive and roughly 8 out of 10 of those infected are now on ART (2). Therefore, HIV and ART may be contributing to the burden of CVD in Malawi. Currently, there are only a few studies assessing CVD risk in the HIV patient population on ART. In Malawi, no such studies exist. Therefore, the investigators propose a novel study assessing baseline cardiovascular disease risk using two novel ultrasound technologies in HIV patients on ART. Cardiovascular disease risk will be assessed using surrogate cardiovascular markers of disease. These surrogates include markers of endothelial function and cardiovascular modulating inflammatory biomarkers. The inflammatory biomarkers measured will be TNF-alpha, IL-6, and CRP. Aspirin, by way of its antiplatelet and anti-inflammatory effect has been demonstrated to inhibit atherosclerosis by way of decreasing TNF-alpha, IL-6, CRP and improving endothelial function. Therefore a second aim of the study will be to demonstrate that aspirin improves surrogate markers of atherosclerosis.

DETAILED DESCRIPTION:
To address our objectives we have designed a six-month prospective randomized controlled study (RCT) investigating cardiovascular disease risk in HIV patients on ART with the implementation of an aspirin versus placebo strategy to investigate whether this risk can be modified. As nearly all HIV patients are anticipated to be on ART in the upcoming decade, we have decided to open this study to only virally suppressed HIV on ART. A total of 100 virally suppressed HIV positive Malawians on ART will be enrolled in this study. Initial screening will occur in the patient population identified as being HIV positive with viral load suppression on ART in the last 3 months. The initial screening will provide cross-sectional information on baseline demographic, clinical, and laboratory characteristics of virally suppressed HIV patients on ART and will assess baseline cardiovascular risk using laboratory biomarker data and endothelial function as surrogate markers (see section under procedures). Ability of distal arteries to dilate under stress will be measured using novel ultrasound technologies applicable to the limited resource healthcare settings in Malawi. After initial screening, eligibility into the study will be determined and selected participants will be randomized into one of two arms:

1. Oral aspirin 325mg daily
2. Oral placebo daily.

This longitudinal RCT will reassess cardiovascular risk at the one-month, 3-month, and six-month mark using the same CVD surrogate measurements of atherosclerosis performed during the initial screening.

Procedures assessing surrogate CVD markers for atherosclerosis:

1. Laboratory analysis (Venipuncture): Inflammatory biomarkers

   • C-Reactive Protein (CRP), Interleukin-6, Tumor Necrosis Factor- alpha
2. Endo-PAT analysis
3. Brachial Flow Mediated dilation
4. Carotid Intima-Media Thickness

ELIGIBILITY:
Inclusion Criteria:

Malawian men and women ages 18-70 who are HIV positive and on ART for at least 6 months on standard therapy (1st line, 2nd line or 3rd line). The HIV viral load at time of enrollment must be suppressed confirmed by HIV DNA PCR in the last 60 days.

Exclusion Criteria:

All patients with risk factors that result in endothelial dysfunction and atherosclerosis will be excluded based on the following exclusion criteria. The rationale behind this is to isolate the effects of virally suppressed HIV on endothelial activity.

1. Presence of HIV viral load in the last 60 days
2. History of diagnosed Diabetes Mellitus
3. Fasting blood sugar >110 at time of enrollment determined by glucose on chemistry profile
4. Uncontrolled Hypertension defined as systolic blood pressure > or equal to 140 and or diastolic >100 mmHg at time of enrollment
5. AST or ALT >200 within the last 30 days. If not obtained in this interval, a baseline AST/ALT will be obtained
6. Renal Failure at time of recruitment (Gfr. <60ml/min/1.73) based on Cockcroft Gault equation.
7. History of myocardial infarction, peripheral vascular disease, cerebrovascular disease. These will also be assessed clinically at the time of enrollment
8. Health condition that would place patient at a health risk for perfusion ischemia during EndoPAT, FMD, CIMT measurement.
9. Current tobacco use or history of tobacco use in the last 90 days
10. Platelet count less than 100 at time of enrollment
11. History of active brain mass/lesion
12. Gastrointestinal bleeding in last 12 months
13. History of hemorrhagic stroke
14. Major life threatening bleeding in the last 12 months
15. Patients considered to be a high bleed risk based on physician assessment
16. History of medication noncompliance in last 3 months
17. Pregnancy
18. Contraindications to aspirin

    * Previous allergic reaction to aspirin or similar medications to aspirin
    * Asthma with nasal congestion or nasal polyps
    * Bleeding disorders (inherited or acquired)
    * Chicken pox

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2015-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Reactive Hyperemia Index | Baseline, 30 days after treatment, 60 days after treatment, 90 days after treatment
  Assessment of peripheral arterial endothelial function
Quantification of inflammatory biomarkers- TNF-alpha, C-Reactive Protein, Interleukin-6 | Baseline, 30 days after treatment, 60 days after treatment, 90 days after treatment.
  Assessment of biochemical surrogates of cardiovascular disease

SECONDARY OUTCOMES:
Bleeding | 30 days, 60 days, 90 days.
Hemoglobin | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anil Purohit, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Lighthouse Trust, Lilongwe, Malawi